CLINICAL TRIAL: NCT07043595
Title: Neuronal Mechanisms Underlying H-Reflex Suppression During Mechanical Loading: The Role of Bone Myoregulation Reflex in Standing Humans
Brief Title: H-Reflex Suppression by Bone Myoregulation Reflex During Mechanical Loading in Standing Humans
Acronym: BMR-HREF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Selim Sezikli, Specialist in Physical Medicine and Rehabilitation, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HReflexBMR2025
Record Dates: First submitted 2025-06-22; First posted 2025-06-29 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: H-reflex; Spinal Reflexes; Posture; Weight-Bearing; Neuromuscular Physiology
Keywords: Bone Myoregulation Reflex; Whole-Body Vibration; Electrophysiology; Soleus Muscle; Presynaptic Inhibition; Mechanoreceptors; Reflex Suppression

STUDY DESIGN:
Intervention Model Description: Single-group crossover design in which each participant undergoes all experimental conditions in a fixed order, including quiet standing, weight-shifting, and whole-body vibration. Electrophysiological recordings are obtained during each condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postural Loading and Vibration Arm (Experimental): Participants in this arm will undergo a sequence of experimental conditions involving postural and mechanical loading. The protocol includes standing quietly on both feet, standing on one foot (right or left), and standing during whole-body vibration (WBV). H-reflex recordings will be obtained from the soleus muscle during each condition to assess changes in spinal reflex excitability.
  Interventions: Procedure: Whole-Body Vibration (WBV)

INTERVENTIONS:
Procedure: Whole-Body Vibration (WBV) — Participants will stand quietly in an upright position while whole-body vibration (WBV) is applied through a vibration platform. The vibration stimulus is delivered while the participant's left foot remains on the vibration surface and the right foot is elevated or isolated. H-reflex recordings are taken from the soleus muscle during the procedure to assess spinal reflex modulation due to mechanical loading.
  Other Names: WBV

SUMMARY:
This study aims to investigate how standing posture and mechanical loading affect reflex responses in the lower limb. Specifically, it focuses on the H-reflex-a type of spinal cord reflex-and how it changes during quiet standing and whole-body vibration. Ten healthy adult volunteers will participate. Researchers will record electrical responses from the calf muscle (soleus) while participants stand still or are exposed to gentle vibration. The goal is to better understand how the nervous system and skeletal system interact in regulating balance and movement.

DETAILED DESCRIPTION:
This study investigates the neural mechanisms responsible for suppression of the H-reflex-a spinal monosynaptic reflex-during mechanical loading in the standing position. Previous research has shown that H-reflex amplitude decreases with increasing postural demand, such as during walking or standing compared to lying down. One hypothesis suggests that this suppression may be mediated not only by vestibular and cutaneous afferents, but also by a bone-derived reflex mechanism called the Bone Myoregulation Reflex (BMR).

In this study, 10 healthy adult volunteers will undergo H-reflex measurements while standing in various loading conditions, including quiet standing and during whole-body vibration (WBV). Participants will stand with one foot isolated from vibration while the other foot is on a vibrating platform. H-reflexes will be recorded from the soleus muscle using standard surface electromyography.

The primary aim is to determine whether BMR contributes to H-reflex suppression during loading. The findings may provide insight into the interaction between skeletal loading and spinal reflex modulation, with potential relevance to balance, gait, and rehabilitation science.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 20 to 45 years
* Able to stand independently for at least 10 minutes
* No known neurological, orthopedic, or balance disorders
* Willingness to participate and provide informed consent

Exclusion Criteria:

* History of spinal cord injury, peripheral neuropathy, or muscle disease
* Recent lower limb surgery or musculoskeletal trauma
* Current use of medications affecting neuromuscular function
* Pregnancy
* Any contraindications to exposure to mechanical vibration

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2025-06-24 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
H-reflex Amplitude | Day 1 (single-session, during each experimental condition)
  The amplitude of the H-reflex recorded from the soleus muscle, evoked at 15% Mmax stimulation level, will be measured during each condition (quiet standing, one-leg stance, and whole-body vibration). The primary aim is to assess changes in spinal excitability due to mechanical loading.

SECONDARY OUTCOMES:
Background EMG Activity | Day 1 (450 ms window prior to stimulation)
  Background electromyographic activity of the soleus muscle will be evaluated over a 450 ms window prior to stimulation to ensure muscle quiescence and verify that changes in reflex amplitude are not due to background activity.

CONTACTS AND LOCATIONS:
Overall Officials: Selim Sezikli, MD, Principal Investigator — Istanbul Physical Medicine and Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the small sample size and the nature of the study, which focuses on basic physiological measurements in healthy volunteers. No data repository is currently planned.